CLINICAL TRIAL: NCT04098289
Title: Effect of Hysteroscopic Septum Resection on Preterm Birth Rate in Singleton Pregnancies After Primary Infertility Treatment
Brief Title: Preterm Delivery After Septum Resection
Acronym: PLEASURE-1
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: PLEASURE-1
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Septum; Uterus; Infertility, Female; Preterm Birth
Keywords: Hysteroscopy; Metroplasty; Primary infertility; Preterm delivery
MeSH Terms: conditions — Infertility, Female; Premature Birth | interventions — Fertilization in Vitro

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hysteroscopic septum resection without in vitro fertilization: Primary infertile women who underwent hysteroscopic septum resection and obtained the first pregnancy with natural conception (without the use of in vitro fertilization techniques).
  Interventions: Procedure: Hysteroscopic septum resection
- Hysteroscopic septum resection with in vitro fertilization: Primary infertile women who underwent hysteroscopic septum resection and obtained the first pregnancy with the use of in vitro fertilization techniques.
  Interventions: Procedure: Hysteroscopic septum resection; Procedure: In vitro fertilization
- Natural conception, without hysteroscopic septum resection: Primary infertile women who did not undergo hysteroscopic septum resection and obtained the first pregnancy with natural conception (without in vitro fertilization techniques).
- In vitro fertilization, without hysteroscopic septum resection: Primary infertile women who did not undergo hysteroscopic septum resection and obtained the first pregnancy with the use of in vitro fertilization techniques.
  Interventions: Procedure: In vitro fertilization

INTERVENTIONS:
Procedure: Hysteroscopic septum resection — Hysteroscopic septum resection, using a 26 French continuous-flow resectoscope with monopolar energy and electrolyte-free distension medium.
  Groups: Hysteroscopic septum resection with in vitro fertilization; Hysteroscopic septum resection without in vitro fertilization
Procedure: In vitro fertilization — Fertilization of oocytes with the spermatozoa of the partner, after induction of ovulation and capacitation of the sperm, using fertilization in vitro and embryo transfer (FIVET) or intracytoplasmic sperm injection (ICSI).
  Groups: Hysteroscopic septum resection with in vitro fertilization; In vitro fertilization, without hysteroscopic septum resection

SUMMARY:
Uterine septum is the most common congenital uterine malformation. It accounts for approximately 35% of all uterine malformations, while the frequency of uterine malformations in the general fertile population is estimated to be between 1% and 4%.

The presence of a uterine septum is associated with subfertility and a high incidence of obstetric complications, such as spontaneous abortion, 3-fold increase in preterm premature rupture of the membranes (PROM), 6-fold increase in preterm delivery, malpresentation at delivery, caesarean section, and increased perinatal morbidity and mortality.

Some studies have found that surgical resection of the uterine septum improves pregnancy outcomes and significantly reduces the risk of preterm delivery. Therefore, the risk for a short-term adverse outcome and long-term sequelae due to preterm delivery such as intraventricular hemorrhage, necrotizing enterocolitis, sepsis, patent ductus arteriosus, retinopathy, deafness, chronic lung disease, cerebral palsy, perinatal death, and impaired mental development in women with uterine septum could be lowered by performing a relatively simple and safe hysteroscopic septum resection (HSR).

However, there are two major concerns regarding HSR: cervical incompetence due to excessive dilatation during hysteroscopy and the rare yet serious complication of uterine rupture in subsequent pregnancy or delivery.

Considering these elements, the aim of this study will be to evaluate the rate of preterm delivery in singleton pregnancy comparing primary infertile women who underwent HSR and who did not undergo the same procedure, with our without in vitro fertilization.

ELIGIBILITY:
Inclusion Criteria:

* Female primary infertility
* Singleton pregnancies

Exclusion Criteria:

* Female secondary infertility
* Multiple pregnancies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women affected by primary infertility who obtained the first ongoing pregnancy with (cases) or without (controls) previous hysteroscopic septum resection, with or without in vitro fertilization.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Preterm delivery rate | Through study completion, an average of 5 year
  Percentage of delivery that occurs before the start of the 37th week of pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Ban Frangež, M.D., Study Director — University of Ljubljana; Jana Miklavcic, M.D., Principal Investigator — University of Ljubljana; Antonio Simone Laganà, M.D., Study Chair — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided